CLINICAL TRIAL: NCT05923593
Title: Tolerance and Safety of an Oral Nutritional Supplement Containing Monoacylglycerol Oil (MAG Oil) as the Main Lipid Source in Healthy Adolescents
Brief Title: Tolerance and Safety of an Oral Nutritional Supplement (Adolescent Cohort)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2214NR
Record Dates: First submitted 2023-02-27; First posted 2023-06-28 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral nutritional supplement (Experimental): Oral nutritional supplement that contains MAG oil
  Interventions: Dietary Supplement: MAG oil oral nutritional supplement (ONS)

INTERVENTIONS:
Dietary Supplement: MAG oil oral nutritional supplement (ONS) — The study product is suitable for use as an oral nutritional supplement (ONS).The study product contains MAG oil.

SUMMARY:
This is an open label, non-randomized, interventional, single arm study.

DETAILED DESCRIPTION:
The primary objective is to assess whether the MAG oil-containing study formula is well tolerated and safe when used as an ONS in healthy adolescents.

Hypothesis: The study product will be safe and well tolerated in healthy adolescents (as previously observed in adults).

Secondary objectives:

1. Describe the frequency and characteristics of possible gastrointestinal intolerance symptoms
2. Describe stool characteristics specifically stool frequency and consistency
3. Describe changes in anthropometric parameters, particularly weight and body mass index (BMI)
4. Describe changes in blood parameters of lipid metabolism
5. Describe changes in hematological and serum biochemistry parameters
6. Describe daily ONS intake and overall compliance

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged 12-17 years
2. BMI range between the 10th and 90th percentile according to the Swiss growth charts with a minimum body weight of 40 kg.
3. Deemed able to comply with study protocol for the study period
4. Able to obtain written informed consent from participants and legally authorized representative(s)

Exclusion Criteria:

1. Pre-existing chronic medical or psychiatric conditions.
2. History of a chronic gastrointestinal disorder (e.g., inflammatory bowel disease, irritable bowel syndrome, celiac disease etc.), or chronic or recurrent gastrointestinal symptoms, including self-reported symptoms such as abdominal pain.
3. Recent episode of an acute gastrointestinal illness with significant gastrointestinal symptoms in the 7 days prior to enrolment.
4. History of chronic constipation (with passage of fewer than 3 spontaneous bowel movements per week on average or history of painful or hard bowel movements), OR chronic or intermittent diarrhea with loose or watery bowel movements ≥ 3 times per day.
5. Colonoscopy or other bowel cleansing procedures within 4 weeks prior to enrolment.
6. Prior use of prescription medication(s), in particular antibiotics, antiacids, laxatives, antidiarrheal agents or other medications impacting gastrointestinal transit time, within 3 weeks prior to enrolment.
7. Significant medical or surgical event in the past 3 months potentially interfering with study procedures and assessments.
8. Subjects following a weight loss program including a low-carbohydrate or low-fat diet, ketogenic diet, intermittent fasting, or any other special diet.
9. Known food allergy in particular cow's milk protein allergy or known/suspected hypersensitivity or intolerance to any other ingredients in the study product. Subjects experiencing gastrointestinal symptoms when consuming dairy products or avoiding dairy in their diet should not participate in the study.
10. Subjects taking energy or protein supplements.
11. Known alcohol or substance abuse.
12. Pregnant or lactating females or having given birth in the past 6 months prior to enrolment. Pregnancy will be ruled out by performing a standard urine dipstick test to female participants of childbearing potential prior to enrolment.
13. Family or hierarchical relationships with Clinical Innovation Lab staff

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects who develop significant gastrointestinal adverse events (deemed probably related or related to study product as per investigator's opinion) leading to discontinuation of the study product and withdrawal from the study | Day 2 to Day 15
  Number of subjects who develop significant gastrointestinal adverse events leading to discontinuation of the study product and withdrawal from the study

SECONDARY OUTCOMES:
Severity of gastrointestinal intolerance symptoms | Day 1 to Day 15
  Individual gastrointestinal symptom scores assessed by the Visual Analogue Scale (VAS) tool from 0 (no symptom) to 10 (maximum severity)
Severity of gastrointestinal intolerance symptoms | Day 1 and Day 15
  Individual gastrointestinal symptom scores assessed by the Gastrointestinal Symptom Rating Scale (GSRS) questionnaire from No discomfort at all (no discomfort) to Very severe discomfort (maximum discomfort)
Change in stool frequency | Day 1 to Day 15
  Assessed by a questionnaire on daily number of stools
Change in stool consistency | Day 1 to Day 15
  Assessed by Bristol Stool Scale from stool consistency A (Separate hard lumps, like nuts, hard to pass) to G (Watery, no solid pieces)
Change in weight | Day 1 and Day 15
  Measured with a weight scale
Change in BMI | Day 1 and Day 15
  Measured with a weight scale and size scale
Changes in lipid profile in the blood | Day 1 and Day 15
  Triglycerides, cholesterol (total cholesterol, LDL cholesterol and HDL cholesterol) measured in plasma
Changes in liver function tests in the blood | Day 1 and Day 15
  ALAT measured in plasma
Changes in liver function tests in the blood | Day 1 and Day 15
  ASAT measured in plasma
Changes in liver function tests in the blood | Day 1 and Day 15
  phosphatase alkaline measured in plasma
Changes in liver function tests in the blood | Day 1 and Day 15
  Gamma glutamyl transferase measured in plasma
Changes in liver function tests in the blood | Day 1 and Day 15
  Total and direct bilirubin measured in plasma
Changes in liver function tests in the blood | Day 1 and Day 15
  Protein and albumin measured in plasma
Changes in renal function tests in the blood | Day 1 and Day 15
  Urea, creatinine measured in plasma
Changes in blood chemistry tests | Day 1 and Day 15
  C-Reactive Protein measured in serum
Changes in blood chemistry tests | Day 1 and Day 15
  Glucose measured in serum
Changes in blood chemistry tests | Day 1 and Day 15
  Sodium measured in serum
Changes in blood chemistry tests | Day 1 and Day 15
  Potassium measured in serum
Changes in blood chemistry tests | Day 1 and Day 15
  Calcium measured in serum
Changes in blood chemistry tests | Day 1 and Day 15
  Phosphate measured in serum
Changes in blood chemistry tests | Day 1 and Day 15
  Magnesium measured in serum
Changes in blood chemistry tests | Day 1 and Day 15
  Chloride measured in serum
Daily intake of study product | Day 1 to Day 15
  Number of participants adhering to daily intake of the study product assessed by a daily questionnaire
Changes in full blood count | Day 1 and Day 15
  thrombocyte count
Changes in full blood count | Day 1 and Day 15
  Erythrocyte count
Changes in full blood count | Day 1 and Day 15
  haemoglobin measured in blood
Changes in full blood count | Day 1 and Day 15
  haematocrit measured in blood
Changes in full blood count | Day 1 and Day 15
  mean cell hemoglobin concentation measured in Blood
Changes in fatty acids profile | Day 1 and Day 15
  Plasma and erythrocytes fatty acids profile
Change in Vitamin A level | Day 1 and Day 15
  Change in serum Vitamin A
Change in 25-hydroxy vitamin D level | Day 1 and Day 15
  Change in serum 25-hydroxy vitamin D
Change in vitamin E level | Day 1 and Day 15
  Change in serum vitamin E
Changes in Vitamin K level | Day 1 and Day 15
  change in international normalized ratio
Changes in in fat-soluble vitamins | Day 1 and Day 15
  Vitamin E/cholesterol ratio measured in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Sun, Principal Investigator — Neslté
Locations (1):
- Clinical Innovation Lab., Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zemrani B, Krattinger LF, Giuffrida F, Corthesy J, Ran-Ressler RR, Benyacoub J. Safety and tolerability of Monoacylglycerol-rich oil as a novel predigested dietary fat source of an enteral formula in healthy adults and adolescents: Two single-arm, open-label studies. Clin Nutr ESPEN. 2025 Feb;65:339-347. doi: 10.1016/j.clnesp.2024.12.014. Epub 2024 Dec 15. PMID 39681164